CLINICAL TRIAL: NCT07162987
Title: Prehabilitation to Patients With Prostate Cancer, Who Are About to Receive Androgen Deprivation Therapy and Radiation Therapy
Brief Title: Prehabilitation to Patients With Prostate Cancer
Acronym: PREPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: REHPA, The Danish Knowledge Centre for Rehabilitation and Palliative Care (Other); Vejle Hospital (Other); Esbjerg Municipality (Other Government); Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25/31257
Record Dates: First submitted 2025-07-30; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer (Diagnosis)
Keywords: prostate cancer; prehabilitation; androgen deprivation therapy; radiation therapy
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving prehabilitation (Experimental): The prehabilitation intervention includes: - Education about the disease and treatment - Physical exsercise training - Values in life - Energy preservation - Nutrition with a focus on hormone therapy - Identiy and role changes - Intimacy and sexuality - Sleep - Pelvic floor training - An individual session with a healthcare professional incl. goal setting
  Interventions: Behavioral: Prehabilitation

INTERVENTIONS:
Behavioral: Prehabilitation — Please refer to arm description

SUMMARY:
The goal of this feasibility study is to test a newly developed, multicomponent prehabilitation intervention to patients with prostate cancer, to improve their resilience to treatment side-effects. The main questions it aims to answer are:

* Are patients and their close relatives willing to take part in prehabilitation?
* What is the acceptability and feasibility of the prehabilitation intervention, seen from the perspectives of patients, their close relatives, and healthcare professionals?
* Are the planned data collection methods feasible, and are there indications of a clinical effect?

Participants will:

* Take part in 12 weeks of physical exercise training
* Attend a 4-day residential prehabilitation intervention, where they receive education and do exercises. After 12 weeks, it is possible to take part in a voluntary follow-up session.
* Patients will respond to questionnaires about their health, symptoms, and quality of life. Patients and their close relatives will attend a group interview. Patients will also complete an exercise diary and brief physical tests

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer
* min 18 years old
* Treatment: Androgen deprivation therapy and raditation therapy
* Resident in Vejle Municipality or Esbjerg Municipality
* Can take part in residential prehabiliation in week 43 or 50, 2025, as well as physical exsercise training in the municipality
* Willing to take part in a research study
* Suited to take part in group sessions
* Be able to read and be understood in Danish
* Be responsible for own personal hygiene and medications at the 4-day residential stay

Exclusion Criteria:

* Persons who do not fulfil the inclusion criteria will be excluded

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to follow-up in quality of life measured by EORTC-QLQ-C30 | From baseline (shortly after enrollment) to 24 and 48 weeks later.
  This is a pilot study with one arm only, thus the aim is mainly to test the feasibility of the chosen primary outcome measure, including whether there are tendencies in data that support the aim of participants maintaining stable quality of life. Hence, measured by the European Organization for the Research and Treatment of Cancer Qality of life Questionnaire (EORTC QLQ-C30), the target is unchanged (stable) quality of life measured from baseline to follow-up at 24 and 48 weeks.

SECONDARY OUTCOMES:
Change in prostate-cancer related symptoms and problems from baseline to follow-up measured by the EPIC-26 | Measured at baseline (shortly after recruitment) and at 24 and 48 weeks.
  As with the primary outcome measure, the purpose in this pilot study is mainly to test the feasibility of the chosen secondary outcome measures. One of the secondary outcomes is prostate cancer related quality of life, measured by five domains in the Expanded Prostate Cancer Index Composite (EPIC-26): urinary incontinence (four items), urinary irritation/obstruction (four items), bowel (six items), sexual (six items) and vitality/hormonal function (five items) and a single-item measure of overall urinary bother. The aim is for the scores in these domains to remain stable from baseline to follow-up at 24 and 48 weeks.
Change in fatigue from baseline to follow-up using the BFI | Measured at baseline (shortly after inclusion) and at 24 and 48 weeks.
  Measured by the Brief Fatigue Inventory (BFI), the aim is stable levels of fatigue from baseline to follow-up at 24 and 48 weeks.
Change in anxiety from baseline to follow up measured by the GAD-7 | At baseline (shortly after inclusion) and at 24 and 48 weeks.
  As with all other measures tested in this one-armed pilot study, the main aim is to test the feasibility of the chosen outcome measures.
  We aim to measure change in anxiety from baseline to follow-up at 24 and 48 weeks measured by the Generalized Anxiety Disorder 7-item (GAD-7) questionnaire. The target is unchanged anxiety.
Change in depression from baseline to follow-up measured by the PHQ-9 | Measured at baseline (shortly after inclusion) and at 24 and 48 weeks
  We aim to measure depression severity using the Patient Health Questionnaire-9 (PHQ-9). The target is unchanged depression score from baseline to follow-up.
Change in BMI from baseline to follow-up calculated from self-reported height and weight | Baseline and at 24 and 48 weeks.
  Change in body mass index (BMI) can be calculated after retrieving the patients' weight and height. Height in meters will be collected at baseline by self-report (through a patient questionnaire). Weight in kilograms will be collected at baseline and follow-up also by self-report. Weight and height will hereafter be combined to report BMI in kg/m^2. The target is no change in BMI from baseline to follow-up.
Change in muscle strength from baseline to follow-up measured by 30 sec sit-to-stand test | Baseline and after finished exercise training at 12 weeks
  Lower limb muscle strength is measured by the 30 seconds sit-to-stand test. The target is unchanged muscle strength from baseline to follow-up.
Change in function from baseline to follow-up measured by the 6MWT | Baseline and after finished exercise training at 12 weeks
  Functional exercise capacity is measured by the 6-minute walk test (6MWT). The target is no change in functional exercise capacity from baseline to follow-up.

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Esbjerg Hospital, Esbjerg, Region Syddanmark
  - REHPA, the Danish Knowledge Centre for Rehabilitation and Palliative Care, Nyborg, Region Syddanmark
  - Vejle Hospital, Vejle, Region Syddanmark

IPD SHARING:
Plan to Share IPD: Undecided
A de-identified copy of data may be made available to external researchers upon reasonable request.